CLINICAL TRIAL: NCT00508053
Title: When Closing Midline Incisions, do Small Stitches Reduce the Risk for Incisional Hernia, Wound Infection or Dehiscence?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sundsvall Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2-Millbourn
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Last update posted 2007-07-30 (Estimated); Status verified 2007-07

CONDITIONS: Wound Infection; Incisional Hernia; Wound Dehiscence
Keywords: wound infection; incisional hernia; wound dehiscence; wound healing; postoperative complications; surgical techniques
MeSH Terms: conditions — Wound Infection; Incisional Hernia; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Mass closure
  Interventions: Procedure: Mass closure
- 2 (Experimental): Small stitches
  Interventions: Procedure: Small stitches

INTERVENTIONS:
Procedure: Small stitches
  Arms: 2
Procedure: Mass closure
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether a technique using very small stitches when closing a midline incision can reduce the risk for wound complications such as incisional hernia, infection or dehiscence.

DETAILED DESCRIPTION:
Most abdominal surgical operations are made through a midline incision and 10% of the patients may get a wound infection. Infection is a risk factor for incisional hernia, which 12 months after the operation can be seen in 10-20% of the patients. Wound dehiscence is seen in approximately 1% of the patients. Surgery because of incisional hernias are common and in Sweden approximately 2000 patients per year needs an operation creating big costs. We know that a midline incision should be closed using a continuous technique, with a suture length to wound length ratio over 4. An earlier interventional study at the Surgical Department in Sundsvall showed that using that technique reduced the risk for hernia with 50%. Subsequent experimental studies indicates that the suture length to wound length ratio should be obtained by small stitches, placed close to each other only incorporating the aponeurosis, and not by large stitches incorporating the complete abdominal wall (mass closure). The hypothesis that midline incisions should be closed with small stitches only incorporating the aponeurosis has to be tested in a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient with an acute or planned operation trough a midline incision at the Surgical Department in Sundsvall, Sweden

Exclusion Criteria:

* Age under 18
* Previous surgery through a midline incision
* Scars from previous surgery crossing the midline
* Preexisting hernia in the midline (umbilical, epigastric)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 737 (Actual)
Dates: Start 2001-01; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Frequency of wound infection | Within the first 30 days after surgery
Frequency of incisional hernia | One year after surgery

SECONDARY OUTCOMES:
Frequency of wound dehiscence | Within the first 10 days after surgery
Effect of different suture techniques on wound complications related to patient characteristics such as age, BMI, sex etc. and operative characteristics such as emergency surgery, type of surgery, degree of contamination, surgeon,etc.. | Within 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Millbourn, MD, Principal Investigator — Sundsvall Hospital
Locations (1):
- Sundsvall Hospital, 851 86 Sundsvall, Sweden

REFERENCES:
- [Derived] Millbourn D, Cengiz Y, Israelsson LA. Effect of stitch length on wound complications after closure of midline incisions: a randomized controlled trial. Arch Surg. 2009 Nov;144(11):1056-9. doi: 10.1001/archsurg.2009.189. PMID 19917943